CLINICAL TRIAL: NCT01987414
Title: Efficacy of a Forearm Rotation Orthosis for Persons With a Hemiparetic Arm
Brief Title: Forearm Rotation Orthosis for Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1309M42881
Record Dates: First submitted 2013-10-29; First posted 2013-11-19 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Stroke
Keywords: Stroke; Cardiovascular Accident; Task-oriented approach; Orthosis; occupational therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Forearm rotation orthosis (6 weeks); Forearm rotation orthosis plus occupational therapy task-oriented approach (6 weeks)
  Interventions: Behavioral: occupational therapy task-oriented approach; Device: Forearm rotation orthosis
- Group B (Active Comparator): no treatment (6 weeks); occupational therapy task-oriented approach (6 weeks)
  Interventions: Behavioral: occupational therapy task-oriented approach; Other: No treatment

INTERVENTIONS:
Behavioral: occupational therapy task-oriented approach — It is a standard treatment in occupational therapy for persons post-stroke or other neurological conditions. It is an approach that emphasizes client-centered, goal-directed, and functional training for restoration of life roles.
  Other Names: OT task-oriented approach
Device: Forearm rotation orthosis — The forearm rotation orthosis is made of Latex-free material and is a custom-molded orthosis designed to assist forearm rotation without limiting functional elbow flexion and extension.
  Arms: Group A
Other: No treatment — Participants will maintain their daily routines during the no treatment period.
  Other Names: control
  Arms: Group B

SUMMARY:
The purpose of this study is to examine the efficacy of a forearm rotation orthosis combined with the occupational therapy task-oriented approach on functional performance for persons with a hemiparetic arm.

Hypotheses of this study are:

1. participants who wear the forearm rotation orthosis will demonstrate significantly greater improvement in functional performance and active range of motion of forearm rotators compared to those who do not;
2. all participants who receive the occupational therapy task-oriented approach intervention will demonstrate significant improvement in functional performance; and
3. all participants who receive the occupational therapy task-oriented approach intervention will demonstrate improvement in motor function of the upper extremity.

DETAILED DESCRIPTION:
Persons with central nervous system (CNS) dysfunction often have difficulty incorporating their affected limb effectively and efficiently into functional tasks due to muscle weakness and/or spasticity. This may further interfere with their performance of everyday activities and restrict life roles. Traditional rehabilitation interventions emphasize spasticity reduction. However, active movement and muscle strength of forearm supination are found strongly related to motor function, rather than spasticity. In contrast, task-oriented movement training trials have demonstrated promising evidence that persons with CNS dysfunction benefit from the training in improvement of motor function and increase functional use of the affected limb.

Orthotic intervention is one therapeutic option for this population. Most orthotic designs for this population are static, developed for sympton reduction or deformity prevention, and aimed at the wrist and hand. However, its effects on spasticity reduction remain controversial. Given that static orthotics may interfere with functional performance and further develop the learned nonuse of the affected limb, a dynamic or mobilization orthosis would be appropriate for enhancing functional performance. Moreover, an orthosis that assists forearm rotation is speculated to enhance functional performance. This study will examine the efficacy of a forearm rotation orthosis combined with the occupational therapy task-oriented approach on functional performance for persons with a hemiparetic arm.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of stroke for at least three months
* Be 18 years of age or older
* Have sufficient cognitive function to follow three-step verbal instruction and provide independent consent
* Have appropriate trunk and lower extremity function that does not interfere with performance of the upper extremity
* Have at least minimum voluntary movement in the upper extremity (10 degrees of shoulder flex/ abduction, 10 degrees of elbow flexion/extension)
* Not receive any rehabilitative interventions concurrent with the study

Exclusion Criteria:

* Severe joint deformities or contractures of the affected upper extremity that limit range of motion required for functional tasks
* Capability of voluntarily extending the wrist and fingers through the full range
* Other rehabilitation interventions concurrent with the study
* Have serious uncontrolled medical problems, such as seizures and visual impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Huang Yu, MS, Principal Investigator — Rehabilitation Science Program at the University of Minnesota; Virgil Mathiowetz, PhD, Study Director — Program in Occupational Therapy, University of Minnesota
Locations (1):
- Children's Rehabilitation Building, University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Information gathered from outcome measures will be shared with other researchers at request. Study PI will seek approval from IRB at the University of Minnesota for means of sharing. Researchers will need to contact the study PI to obtain the information.

REFERENCES:
- [Background] Braendvik SM, Elvrum AK, Vereijken B, Roeleveld K. Relationship between neuromuscular body functions and upper extremity activity in children with cerebral palsy. Dev Med Child Neurol. 2010 Feb;52(2):e29-34. doi: 10.1111/j.1469-8749.2009.03490.x. Epub 2009 Oct 7. PMID 19811515
- [Background] O'Dwyer NJ, Ada L, Neilson PD. Spasticity and muscle contracture following stroke. Brain. 1996 Oct;119 ( Pt 5):1737-49. doi: 10.1093/brain/119.5.1737. PMID 8931594
- [Background] Dunning K, Berberich A, Albers B, Mortellite K, Levine PG, Hill Hermann VA, Page SJ. A four-week, task-specific neuroprosthesis program for a person with no active wrist or finger movement because of chronic stroke. Phys Ther. 2008 Mar;88(3):397-405. doi: 10.2522/ptj.20070087. Epub 2008 Jan 10. PMID 18187493
- [Background] Page SJ, Levine P, Leonard AC. Modified constraint-induced therapy in acute stroke: a randomized controlled pilot study. Neurorehabil Neural Repair. 2005 Mar;19(1):27-32. doi: 10.1177/1545968304272701. PMID 15673841
- [Background] Page SJ, Levine P, Leonard A, Szaflarski JP, Kissela BM. Modified constraint-induced therapy in chronic stroke: results of a single-blinded randomized controlled trial. Phys Ther. 2008 Mar;88(3):333-40. doi: 10.2522/ptj.20060029. Epub 2008 Jan 3. PMID 18174447
- [Background] Taub E, Uswatte G, King DK, Morris D, Crago JE, Chatterjee A. A placebo-controlled trial of constraint-induced movement therapy for upper extremity after stroke. Stroke. 2006 Apr;37(4):1045-9. doi: 10.1161/01.STR.0000206463.66461.97. Epub 2006 Mar 2. PMID 16514097
- [Background] Watanabe T. The role of therapy in spasticity management. Am J Phys Med Rehabil. 2004 Oct;83(10 Suppl):S45-9. doi: 10.1097/01.phm.0000141130.58285.da. PMID 15448577
- [Background] Lannin NA, Horsley SA, Herbert R, McCluskey A, Cusick A. Splinting the hand in the functional position after brain impairment: a randomized, controlled trial. Arch Phys Med Rehabil. 2003 Feb;84(2):297-302. doi: 10.1053/apmr.2003.50031. PMID 12601664
- [Background] Taub E, Uswatte G, Elbert T. New treatments in neurorehabilitation founded on basic research. Nat Rev Neurosci. 2002 Mar;3(3):228-36. doi: 10.1038/nrn754. PMID 11994754
- [Background] Gillen G. Upper extremity function and management. In G. Gillen (Ed.), Stroke rehabilitation: A function-based approach (3rd ed., pp. 218-279). St. Louis: Mosby, 2011.
- [Background] Milazzo S, Gillen G. Splinting applications. In G Gillen (Ed.), Stroke rehabilitation: A function-based approach (3rd ed., pp. 326-349). St. Louis: Mosby, 2011
- [Background] Wolf SL, Winstein CJ, Miller JP, Thompson PA, Taub E, Uswatte G, Morris D, Blanton S, Nichols-Larsen D, Clark PC. Retention of upper limb function in stroke survivors who have received constraint-induced movement therapy: the EXCITE randomised trial. Lancet Neurol. 2008 Jan;7(1):33-40. doi: 10.1016/S1474-4422(07)70294-6. PMID 18077218

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B
Started | 10 | 8
Completed | 8 | 6
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 5 | 13
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: year] | 53.88 (11.99) | 58.5 (10.17) | 55.86 (11.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Canadian Occupational Performance Measure (COPM) - Performance
Description: Used to evaluate participants' self-perceived functional performance. In this structured interview, participants are asked to select 5 tasks to perform and then rate their perception of how well they are able to complete each task on a scale of 1 (unable to perform) to 10 (able to perform extremely well). Total scores are an mean of individual task scores and also range from 1 (unable to perform tasks) to 5 (able to perform tasks extremely well). Collected data will be used to measure changes within and between groups on self-perceived performance between week 1 and 8, week 1 and 15, as well as week 8 and 15.
Time Frame: Week 1, 8, and 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 6
score on a scale
  Week 1 (Pre-test) | 2.95 (.77) | 3.77 (1.33)
  Week 8 (Post-test 1) | 3.3 (1.21) | 3.43 (1.05)
  Week 15 (Post-test 2) | 5.8 (1.34) | 5.98 (1.53)

2. Primary Outcome: Canadian Occupational Performance Measure (COPM) - Satisfaction
Description: Used to evaluate participants' self-perceived satisfaction with performance. In this structured interview, participants are asked to select 5 tasks to perform and then rate their satisfaction of how well they are able to complete each task on a scale of 1 (unsatisfied) to 10 (completely satisfied). Total scores are an mean of individual task scores and also range from 1 (unsatisfied) to 5 (completely satisfied). Collected data will be used to measure changes within and between groups on self-perceived satisfaction with performance between week 1 and 8, week 1 and 15, as well as week 8 and 15.
Time Frame: Week 1, 8, and 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 6
score on a scale
  Week 1 (Pre-test) | 2.73 (1.11) | 3.17 (1.48)
  Week 8 (Post-test 1) | 3.18 (1.54) | 3.1 (1.18)
  Week 15 (Post-test 2) | 5.93 (1.19) | 5.65 (1.29)

3. Primary Outcome: Wolf Motor Function Test (WMFT) - Time
Description: This test will be used to quantitatively assess participants' motor function of the upper extremity. Participants will be asked to complete 15 tasks, each within a 120-second window. The number of seconds required to complete the task is recorded. If the participant exceeds 120 seconds, no additional time will be added and 120 seconds will be recorded. The total score is calculated as a mean of score (in seconds) from the 15 tasks. Collected data will be used to measure changes within and between groups between week 1 and 8, week 1 and 15, as well as week 8 and 15.
Time Frame: Week 1, 8, and 15
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 6
seconds
  Week 1 (Pre-test) | 66.25 (17.99) | 40.38 (40.45)
  Week 8 (Post-test 1) | 63.25 (14.88) | 39.15 (39.49)
  Week 15 (Post-test 2) | 61.41 (15.57) | 44.65 (39.36)

4. Primary Outcome: Wolf Motor Function Test (WMFT) - Function
Description: This test will be used to quantitatively assess participants' motor function of the upper extremity. Participants will be asked to complete 15 tasks, each within a 120-second window. Participants are scored on their ease of completing each task. Scores range from 1 to 3, with higher scores representing greater ease of task completion. The total score is mean value of the 15 item scores. Collected data will be used to measure changes within and between groups between week 1 and 8, week 1 and 15, as well as week 8 and 15.
Time Frame: Week 1, 8, and 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 6
score on a scale
  Week 1 (Pre-test) | 2.07 (.35) | 2.8 (.94)
  Week 8 (Post-test 1) | 2.16 (.41) | 2.77 (1.33)
  Week 15 (Post-test 2) | 2.16 (.36) | 2.9 (1.33)

5. Primary Outcome: Motor Activity Log (MAL) - Amount of Use
Description: This test is used to measuring participants' actual use of the involved arm in the real world. This interview-style test contains 30 items. Participants are asked how often they use their non-dominant arm/hand to complete each of the 30 tasks. Scores range from 0 (never use non-dominant hand) to 5 (normally use non-dominant hand). The total score is a mean of 30 item scores. Collected data will be used to measure changes within and between groups between week 1 and 8, week 1 and 15, as well as week 8 and 15.
Time Frame: Week 1, 8, and 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 6
score on a scale
  Week 1 (Pre-test) | .46 (.42) | 1.06 (.85)
  Week 8 (Post-test 1) | .56 (.57) | 1.01 (.96)
  Week 15 (Post-test 2) | .81 (.64) | 1.61 (1.22)

6. Primary Outcome: Motor Activity Log (MAL) - How Well
Description: This test is used to measuring participants' actual use of the involved arm in the real world. This interview-style test contains 30 items. Participants are asked how well they use their non-dominant arm/hand to complete each of the 30 tasks. Scores range from 0 (never use non-dominant hand) to 5 (normal use of non-dominant hand). The total score is a mean of 30 item scores. Collected data will be used to measure changes within and between groups between week 1 and 8, week 1 and 15, as well as week 8 and 15.
Time Frame: Week 1, 8, and 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 6
units on a scale
  Week 1 (Pre-test) | .52 (.47) | 1.15 (.75)
  Week 8 (Post-test 1) | .56 (.54) | 1.18 (1.19)
  Week 15 (Post-test 2) | .86 (.66) | 1.63 (1.2)

7. Secondary Outcome: Goniometric Measurements - Shoulder Flexion
Description: A goniometer will be used to measure active and passive range of motion of the upper extremity in degrees. Collected data will be used to measure changes within and between groups between week 1 and 8, week 1 and 15, as well as week 8 and 15.
Time Frame: Week 1, 8, and 15
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 6
degrees
  Week 1 (Pre-test) | 103.5 (30.56) | 99 (41.91)
  Week 8 (Post-test 1) | 92.75 (33.52) | 93 (29.15)
  Week 15 (Post-test 2) | 100.38 (38.06) | 96 (29.5)

8. Secondary Outcome: Goniometric Measurements - Shoulder Abduction
Description: as for outcome 7
Time Frame: Week 1, 8, and 15
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 6
degrees
  Week 1 (Pre-test) | 96 (33.56) | 95.17 (32.33)
  Week 8 (Post-test 1) | 85.75 (25.27) | 87.83 (26.28)
  Week 15 (Post-test 2) | 87.75 (31.35) | 90.33 (27.34)

9. Secondary Outcome: Goniometric Measurements - Elbow Extension
Description: as for outcome 7
Time Frame: Week 1, 8, and 15
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 6
degrees
  Week 1 (Pre-test) | 117.25 (17.52) | 103.67 (33.21)
  Week 8 (Post-test 1) | 113.13 (21.01) | 97.5 (21.36)
  Week 15 (Post-test 2) | 125.25 (10.31) | 119.83 (30.22)

10. Secondary Outcome: Goniometric Measurements - Forearm Pronation
Description: as for outcome 7
Time Frame: Week 1, 8, and 15
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 6
degrees
  Week 1 (Pre-test) | 63.13 (19.14) | 67.67 (16.81)
  Week 8 (Post-test 1) | 61.63 (30.42) | 64 (27.94)
  Week 15 (Post-test 2) | 65.63 (23.37) | 59.17 (18.28)

11. Secondary Outcome: Goniometric Measurements - Forearm Supination
Description: as for outcome 7
Time Frame: Week 1, 8, and 15
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 6
degrees
  Week 1 (Pre-test) | 38 (29.89) | 51.33 (24.87)
  Week 8 (Post-test 1) | 38.13 (29.92) | 47.5 (33.58)
  Week 15 (Post-test 2) | 55.13 (27.48) | 53.33 (27.14)

12. Secondary Outcome: Goniometric Measurements - Wrist Extension
Description: as for outcome 7
Time Frame: Week 1, 8, and 15
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 6
degrees
  Week 1 (Pre-test) | 20.25 (17.5) | 36.67 (19.4)
  Week 8 (Post-test 1) | 23.13 (19.81) | 40.38 (22.71)
  Week 15 (Post-test 2) | 26.25 (21.67) | 39.17 (22.23)

13. Secondary Outcome: Upper Extremity Strength - Shoulder Flexion
Description: A hand-held dynamometer will be used to measure upper extremity strength in pounds. Participants are asked to complete each task 3 times. Reported data is the mean of 3 attempts. Collected data will be used to measure changes within and between groups between week 1 and 8, week 1 and 15, as well as week 8 and 15.
Time Frame: Week 1, 8, and 15
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 6
lbs
  Week 1 (Pre-test) | 14.91 (7.01) | 14.48 (6.99)
  Week 8 (Post-test 1) | 15.13 (5.3) | 18.06 (11.53)
  Week 15 (Post-test 2) | 17.36 (10.08) | 21.13 (15.22)

14. Secondary Outcome: Upper Extremity Strength - Shoulder Abduction
Description: as for outcome 13
Time Frame: Week 1, 8, and 15
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 6
lbs
  Week 1 (Pre-test) | 15.1 (6.24) | 17.82 (10.69)
  Week 8 (Post-test 1) | 15.32 (6.57) | 16.99 (11.73)
  Week 15 (Post-test 2) | 17.65 (9.7) | 18.68 (13.61)

15. Secondary Outcome: Upper Extremity Strength - Elbow Extension
Description: as for outcome 13
Time Frame: Week 1, 8, and 15
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 6
lbs
  Week 1 (Pre-test) | 12.9 (5.27) | 13.97 (7.77)
  Week 8 (Post-test 1) | 11.98 (3.13) | 16.43 (7.81)
  Week 15 (Post-test 2) | 12.81 (6.62) | 17.56 (10.46)

16. Secondary Outcome: Upper Extremity Strength - Forearm Pronation
Description: as for outcome 13
Time Frame: Week 1, 8, and 15
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 6
lbs
  Week 1 (Pre-test) | 10.83 (4.99) | 11.87 (5.49)
  Week 8 (Post-test 1) | 10.97 (3.6) | 11.51 (6.3)
  Week 15 (Post-test 2) | 11.74 (6.29) | 11.98 (9.96)

17. Secondary Outcome: Upper Extremity Strength - Forearm Supination
Description: as for outcome 13
Time Frame: Week 1, 8, and 15
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 6
lbs
  Week 1 (Pre-test) | 6.06 (4.86) | 7.74 (3.74)
  Week 8 (Post-test 1) | 5.76 (3.56) | 6.58 (3.12)
  Week 15 (Post-test 2) | 6.3 (3.36) | 8.15 (3.74)

18. Secondary Outcome: Upper Extremity Strength - Wrist Extension
Description: as for outcome 13
Time Frame: Week 1, 8, and 15
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 6
lbs
  Week 1 (Pre-test) | 8.72 (6.13) | 11.98 (7.2)
  Week 8 (Post-test 1) | 8.38 (5.76) | 15.2 (11.59)
  Week 15 (Post-test 2) | 9.74 (6.17) | 14.79 (11.31)

19. Secondary Outcome: Upper Extremity Strength - Grip
Description: A Jamar Dynamometer will be used to measure grip strength in pounds. Participants are asked to complete this task 3 times. Reported data is the mean of 3 attempts. Collected data will be used to measure changes within and between groups between week 1 and 8, week 1 and 15, as well as week 8 and 15.
Time Frame: Week 1, 8, and 15
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 6
lbs
  Week 1 (Pre-test) | 13.21 (7.06) | 29.39 (18.83)
  Week 8 (Post-test 1) | 13.77 (9.62) | 28.5 (22.33)
  Week 15 (Post-test 2) | 17.38 (6.79) | 28.55 (17.76)

20. Secondary Outcome: Upper Extremity Strength - Palmar Pinch
Description: A pinch gauge will be used to measure pinch strength in pounds. Participants are asked to complete this task 3 times. Reported data is the mean of 3 attempts. Collected data will be used to measure changes within and between groups between week 1 and 8, week 1 and 15, as well as week 8 and 15.
Time Frame: Week 1, 8, and 15
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 6
lbs
  Week 1 (Pre-test) | .67 (1.28) | 6.06 (6.5)
  Week 8 (Post-test 1) | .88 (1.1) | 4.95 (6.71)
  Week 15 (Post-test 2) | 1.17 (1.73) | 5.11 (5.78)

21. Secondary Outcome: Upper Extremity Strength - Lateral Pinch
Description: as for outcome 20
Time Frame: Week 1, 8, and 15
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 6
lbs
  Week 1 (Pre-test) | 6.94 (3.71) | 17.72 (12.61)
  Week 8 (Post-test 1) | 7.32 (4.82) | 16.72 (14.28)
  Week 15 (Post-test 2) | 9.27 (3.53) | 16.84 (11.13)

ADVERSE EVENTS:
Time Frame: 15 weeks
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 0/8 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/14/NCT01987414/Prot_SAP_000.pdf